CLINICAL TRIAL: NCT01975649
Title: Effects of Tribulus Terrestris in Postmenopausal Women With Hypoactive Sexual Desire Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Selmo Geber, MD, PhD, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TTC; 245.553C (Other: COEP)
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Menopause; Sexual Abstinence
Keywords: postmenopausal; hypoactive; sexual disorder; androgen
MeSH Terms: conditions — Sexual Abstinence; Sedentary Behavior; Sexual Dysfunction, Physiological | interventions — Tribulus extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tribulus Terrestris (Experimental): patients will use Tribulus terrestris (750 mg/day) during 120 days
  Interventions: Drug: Tribulus Terrestris
- Placebo (Placebo Comparator): patients will use placebo for 120 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tribulus Terrestris — patients will use 750 mg/day during 120 days
  Other Names: tribulus
  Arms: Tribulus Terrestris
Other: Placebo — patients will use placebo pills with the same shape of the drug
  Arms: Placebo

SUMMARY:
Hypoactive Sexual Desire Disorder ( HSDD ) is very common in postmenopausal women due to a reduction in circulating androgen levels. The aim of this study is to evaluate the effects of Tribulus Terrestris in premenopausal women with HSDD.

DETAILED DESCRIPTION:
Hypoactive Sexual Desire Disorder ( HSDD ) is the most prevalent female sexual dysfunction in society mainly in postmenopausal women, and is strongly linked to the quality of life of women . The androgen hormones decline over age in the premenopausal period, more sharply after menopause. Tribulus terrestris is a plant native to India , recommended in the treatment of infertility , low libido and impotence . Its main active ingredient is the protodioscin , which has been attributed to an increase in testosterone levels and improved sexual function . The aim of this study is to evaluate the effects of Tribulus Terrestris in premenopausal women with HSDD .

ELIGIBILITY:
Inclusion Criteria:

* at least one year after last menstrual period
* with no use of hormonal replacement therapy within the last 3 months
* without any medication, drugs or alcohol.
* Healthy patients without systemic or psychiatric disease

Exclusion Criteria:

* Patient smoker (10 cigarettes per day).
* Patients with blood pressure > 160/90 mm Hg.
* Patient with breast or endometrial carcinoma.
* Patients with a history of myocardial infarction.
* Patient with Diabetes.
* Patient with vaginal bleeding from any source.
* Patients with hepatic injury.
* Patients with active thrombophlebitis or thromboembolic disorders recent
* Patients with interpersonal relationship problems with your relationship or partner
* Patients with sexual problems from your partner

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Sexual Desire | 120 days
  we will use the "Quotient Sexual - Version Feminine (QS-F) brazilian questionary to make the evaluation

SECONDARY OUTCOMES:
serum levels of prolactin and thyroid-stimulating hormone (TSH) | 120 days
  Blood test

OTHER OUTCOMES:
serum levels of testosterone and sex hormone-binding globulin (SHBG) | 120 days
  Blood test

CONTACTS AND LOCATIONS:
Overall Officials: Selmo Geber, MD PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Hospital das Clinicas - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil